CLINICAL TRIAL: NCT07091890
Title: Microbiology and Clinical Efficacy of Professional Topical Fluoride on Streptococcus Mutans and Selemonas Sputigena in Orthodontic Patients: a Randomized Clinical Trial
Brief Title: Effects of Topical Fluoride in Orthodontic Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Alessia Pardo, Principal Investigator, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 328CET
Record Dates: First submitted 2025-07-10; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Topical Fluoride; Orthodontic Patients; Antimicrobial Effect; Clinical Effect

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Professional oral hygiene session and a topical fluoride prophylaxis treatment with gel (Experimental)
  Interventions: Device: Fluoride gel
- Professional oral hygiene session and a topical fluoride prophylaxis treatment with varnish (Experimental)
  Interventions: Device: Fluoride varnish
- Professional oral hygiene session alone (No Intervention): All patients underwent a professional oral hygiene session to remove bacterial plaque and calculus from the tooth surfaces. Bacterial plaque was removed using a supragingival air-polishing device that dispersed glycine powder. When calcified residues were present, a piezoelectric ultrasonic scaler with either a supragingival insert, perio-slim periodontal insert, or scaler was selectively used in cases of deposits in areas that were difficult to access

INTERVENTIONS:
Device: Fluoride gel — After non-surgical therapy, 6-8 g of a gel containing 12,500 ppm of fluoride was applied for 4 min using a disposable tray appropriately sized for the patient's mouth. As per the guidelines, the patient was asked to briefly rinse their mouth with water. The aim was to remineralize the dental enamel to make it less susceptible to acid attacks caused by low salivary pH and the byproducts of bacterial metabolism
  Arms: Professional oral hygiene session and a topical fluoride prophylaxis treatment with gel
Device: Fluoride varnish — After non-surgical therapy, a fluoride varnish containing 7,700 ppm of fluoride in a homogeneous solution was evenly distributed over the dental surfaces using a micro-brush. Patients were instructed to spit out excess saliva but not to rinse their mouth with water, and to refrain from eating or drinking for at least 60 min afterward. After drying, the varnish formed a fluoride-rich layer on the enamel, increasing the concentration by up to four times. Despite the high concentration of fluoride, the resin component of the varnish allowed for a slow, controlled release of fluoride over time, thus preventing its immediate loss and minimizing the amount ingested by the patient. The purpose was to prevent mineral loss from the enamel and promote its restoration, making the dental tissue more resistant to the acidic pH of saliva caused by the production of organic acids through bacterial metabolism.
  Arms: Professional oral hygiene session and a topical fluoride prophylaxis treatment with varnish

SUMMARY:
This study was born from the need to improve caries prevention in orthodontic patients, a group particularly at risk. Fixed orthodontic appliances make daily oral hygiene more difficult, leading to increased plaque accumulation and the proliferation of cariogenic bacteria such as Streptococcus mutans and, more recently, Selenomonas sputigena. Although the latter does not cause cavities on its own, it enhances the action of Streptococcus mutans, making the caries process more aggressive.

The aim of the research was to evaluate the effectiveness of two different types of professional topical fluoride-gel and varnish-in reducing the presence of these bacteria and improving certain clinical parameters, such as salivary pH, the DMFT index (which measures decayed, missing, and filled teeth), and the Plaque Control Record (PCR%).

The study involved 45 patients, all between 8 and 17 years old and wearing fixed orthodontic appliances. They were divided into three groups: one received fluoride gel, another received fluoride varnish, and the third group underwent only a professional oral hygiene session, without any fluoride application. All patients were evaluated at the beginning of the study (T0) and again after four months (T1), both clinically and microbiologically, through saliva and plaque analysis.

The results showed that in the fluoride-treated groups-especially the varnish group-there was a significant reduction in plaque, an improvement in salivary pH (mainly in the gel group), and a decrease in the presence of S. mutans and S. sputigena. Furthermore, there was a reduction in oral Streptococci and Lactobacilli levels in the treated groups, whereas these levels increased in the control group. Interestingly, although not all differences were statistically significant, the improvements observed in the treatment groups suggest a clinically relevant benefit of topical fluoride, especially in varnish form.

In conclusion, professional application of fluoride-whether in gel or varnish form-proved effective in counteracting key bacteria responsible for dental caries in orthodontic patients and in improving several relevant clinical parameters. This confirms the importance of combining professional oral hygiene with specific fluoride treatments in patients wearing orthodontic appliances.

ELIGIBILITY:
Inclusion Criteria:

* 1 < DMFT < n-1 (n= number of teeth present in the oral cavity)
* age between 8 and 17 years
* patient wearing fixed orthodontic appliances

Exclusion Criteria:

* DMFT = 0 *; professional topical fluoride prophylaxis session carried out in the last 3 months
* patient not wearing fixed orthodontic appliances
* orthodontic treatment already completed or not started * DMFT refers to a caries prevalence index related to the presence of Decayed, Missing, Filled Teeth due to caries (Decayed, Missing, Filled Teeth).

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Quantitative evaluation of Streptococcus mutans | T0 baseline, T1 4 months
  Molecular methods Polymerase Chain Reaction - Quantitative Polymerase Chain Reaction (PCR-qPCR)
Quantitative evaluation of Selemonas sputigena | T0 baseline, T1 4 months
  Molecular methods Polymerase Chain Reaction - Quantitative Polymerase Chain Reaction (PCR-qPCR)

SECONDARY OUTCOMES:
Plaque Control Record | T0 baseline, T1 4 months
  The Plaque Control Record (%) indicates the percentage of the tooth surface covered by bacterial plaque. The percentage was calculated by dividing the number of tooth surfaces with plaque by the number of areas examined and then multiplying the result by 100. Four surfaces were examined for each tooth: buccal, lingual/palatal, mesial, and distal surfaces. The highest value is 100% and it means that plaque is present on all the surfaces.
DMFT | T0 baseline, T1 4 months
  The DMFT is a caries prevalence index that refers to the presence of Decayed, Missing, Filled Teeth due to caries (Decayed, Missing, Filled Teeth). The individual value for the patient is the sum of D+M+F. The highest score is 32 and it shows the greatest value for this index.
Salivary ph | T0 baseline, T1 4 months
  To assess salivary pH, a specific pH reagent strip was moistened with the patient's saliva. After an appropriate waiting period, as indicated by the manufacturer of the saliva test, the color displayed by the strip was compared to that on the reference scale to read the result. The scale of pH is: <6,5 acid; 6,5-7,5 neutral; >7,5 alkaline.

CONTACTS AND LOCATIONS:
Locations (1):
- Integrated University Hospital Company Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No